CLINICAL TRIAL: NCT05616234
Title: Exercise-induced Changes in Exosomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1956959
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Exosomes; Connective Tissue; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise trial (Experimental): Participants will perform a bout of exercise. In addition, a baseline and post-exercise blood sample will be drawn.
  Interventions: Procedure: Resistance Exercise

INTERVENTIONS:
Procedure: Resistance Exercise — Participants will perform a bout of lower body resistance exercise consisting of leg press, leg extension and leg curls.

SUMMARY:
The proposed study aims to shed light on the function/importance/relevance of exercise-induced changes in exosomes to connective tissues. Exosomes are known to increase robustly in response to exercise. We have previously shown that serum isolated from subjects after they lift heavy weights increases human engineered ligament collagen content and mechanics more than serum from before they lift weight. Further, we showed that exercise-induced changes in hormones could not explain the change in ligament structure or function. These data indicate that there is a significant gap in our understanding of muscle-connective tissue crosstalk. To address this gap, the current proposal seeks to: i) isolate and sequence exosomal RNA (long non-coding, miR, and mRNA) and ii) determine whether exosomes isolated from serum after exercise increase engineered ligament mechanics and collagen content.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults (18-35 y)
* Experience with exercise (>1y)

Exclusion Criteria:

* Pregnancy
* Smoking
* Receiving any medication that may interfere with the study outcomes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Collagen content of ligament constructs | 15 min post-exercise
  Ligament constructs will be treated for 7 days with experimental feed medium containing serum, or exosomes isolated from serum, obtained at baseline or post-exercise for determination of collagen content using a hydroxyproline assay.

SECONDARY OUTCOMES:
Ultimate tensile stress and modulus of ligament constructs | 15 min post-exercise
  ligament constructs will be treated for 7 days with experimental feed medium containing serum, or exosomes isolated from serum, obtained at baseline or post-exercise for determination of ultimate tensile stress and modulus.
Exosomal RNA | 15 min post-exercise
  Isolation and sequencing of exosomal RNA from serum obtained at baseline or post-exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Hickey Laboratory, Davis, California, United States